CLINICAL TRIAL: NCT05911620
Title: Evaluation of the Severity of Hepatic Fibrosis by Magnetic Resonance Elastography in the Diagnosis of Endogenous Hypercorticism
Acronym: HEPACORT
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Central Hospital, Nancy, France (Other)
Responsible Party: Principal Investigator, SCHEYER Nicolas, Principal Investigator, Central Hospital, Nancy, France
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 2022-A01786-37
Record Dates: First submitted 2023-05-02; First posted 2023-06-22 (Actual); Last update posted 2023-10-25 (Actual); Status verified 2023-10

CONDITIONS: Cushing Syndrome; Metabolic Syndrome
MeSH Terms: conditions — Cushing Syndrome; Metabolic Syndrome | interventions — Elasticity Imaging Techniques

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cushing's Syndrome (Experimental): Patients with proven autonomic cortisol secretion (Cushing's Syndrome)
  Interventions: Device: Magnetic resonance elastography (MRE)
- Suspected Cushing's Syndrome (Experimental): Patients with possible autonomic cortisol secretion (Suspected Cushing's Syndrome)
  Interventions: Device: Magnetic resonance elastography (MRE)
- Metabolic Syndrome (Active Comparator): Patients with metabolic syndrome
  Interventions: Device: Magnetic resonance elastography (MRE)

INTERVENTIONS:
Device: Magnetic resonance elastography (MRE) — Magnetic Resonance Imaging (MRI) imaging with low-frequency vibrations to create a visual map (elastogram) that shows stiffness of body tissues

SUMMARY:
The main hypothesis of the HEPACORT study is that upon diagnosis of endogenous Cushing's syndrome, significant liver fibrosis may be present, particularly in the most severe forms of Cushing's syndrome.

the HEPACORT study is the first exploratory study to assess the severity of liver fibrosis in patients with Cushing's syndrome or suspected of presenting by Magnetic Resonance Elastography (MRE).

ELIGIBILITY:
Inclusion Criteria:

* age ≥ 18 years old;
* Person affiliated to a social security scheme or beneficiary of such a scheme;
* Person having received complete information on the organization of the research and having signed informed consent;
* Person having carried out a preliminary clinical examination adapted to the research.
* Patients with Cushing's syndrome (for the Cushing's Syndrome group)
* Patients with possible Cushing's syndrome (for the suspected Cushing's Syndrome group) defined as response to the dexamethasone supression test with 1 mg of Dexamethasone, with a plasma cortisol assay at 8 am between 18 and 50 µg/L carried out in the 3 months preceding ;
* Patients with metabolic syndrome (for the metabolic syndrome group)

Exclusion Criteria:

* Person having taken corticosteroid therapy for more than 3 months during the 2 years preceding inclusion;
* Person having received corticosteroid therapy of shorter duration with discontinuation less than one month before inclusion;
* Person having taken anticortisolic treatment for more than 3 months during the 2 years preceding inclusion;
* Person with chronic liver disease;
* Person with alcohol misuse, defined by a weekly consumption of more than 10 standard units;
* Person with a morphotype that does not allow an MRI examination to be performed;
* Woman of childbearing age who does not have an effective means of contraception;
* Contraindication to performing an MRI examination.
* Person referred to in Articles L. 1121-5, L. 1121-7 and L1121-8 of the French Public Health Code.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2023-10-24 (Actual); Primary Completion 2026-02-28 (Estimated); Study Completion 2026-08-31 (Estimated)

PRIMARY OUTCOMES:
Estimation of the severity of hepatic fibrosis by MRE (kPa). | Baseline (day 0)
  Estimation of the severity of hepatic fibrosis in kPa by a non-invasive elastography method : magnetic resonance elastography.

SECONDARY OUTCOMES:
Evaluation of the presence of hepatic fibrosis by MRE (kPa). | Baseline (day 0)
  Evaluation of the presence of hepatic fibrosis by ERM : ERM value ≥ 72.5 kPa.
Evaluation of the association between hyperglycemia (blood glucose by g/L) with the presence of Fibrosis by MRE (kPa). | Baseline (day 0)
Evaluation of the association between high blood pressure (mmHg) with the presence of Fibrosis by MRE (kPa). | Baseline (day 0)
Evaluation of the association between overweight (kg) with the presence of Fibrosis by MRE (kPa). | Baseline (day 0)
Evaluation of the association between osteoporosis (g/cm²) with the presence of Fibrosis by MRE (kPa). | Baseline (day 0)
Evolution of transaminases (UI/L) between the diagnosis and the last visit. | 1 year
Evolution of GGT (gamma-glutamyl transferase) (UI/L) between the diagnosis and the last visit. | 1 year
Evolution of ALP (Alkaline Phosphatases) (UI/L) between the diagnosis and the last visit | 1 year
Evolution of Bilirubin (mg/L) between the diagnosis and the last visit. | 1 year
Evolution of Albumin (g/L) between the diagnosis and the last visit. | 1 year
Evolution of platelets (platelets/mm3) between the diagnosis and the last visit. | 1 year
Evolution of ferritin (ng/mL) between the diagnosis and the last visit. | 1 year

CONTACTS AND LOCATIONS:
Locations (1):
- CHRU Nancy, Nancy, France